CLINICAL TRIAL: NCT02223650
Title: A Pilot Randomized Clinical Trial of Overminus Spectacle Therapy for Intermittent Exotropia
Brief Title: A Pilot Clinical Trial of Overminus Spectacle Therapy for Intermittent Exotropia
Acronym: IXT3
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Jaeb Center for Health Research (Other)
Collaborators: Pediatric Eye Disease Investigator Group (Network); National Eye Institute (NEI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IXT3; 2U10EY011751 (NIH)
Record Dates: First submitted 2014-08-20; First posted 2014-08-22 (Estimated); Results first posted 2016-12-20 (Estimated); Last update posted 2017-05-19 (Actual); Status verified 2017-04

CONDITIONS: Intermittent Exotropia
Keywords: Intermittent Exotropia; IXT; overminus

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Overminus Treatment (Experimental): 2.50D overminus spectacles
  Interventions: Device: Overminus treatment
- Non-overminus Treatment (Active Comparator): spectacles without overminus or no spectacles
  Interventions: Device: Non-overminus treatment

INTERVENTIONS:
Device: Overminus treatment — 2.50D overminus spectacles
  Other Names: Overminus spectacles; Overminus glasses; Overminus therapy
  Arms: Overminus Treatment
Device: Non-overminus treatment — spectacles without overminus or no spectacles
  Arms: Non-overminus Treatment

SUMMARY:
The objective of this short-term, pilot randomized trial comparing 2.50 diopters (D) overminus lens treatment vs. non-overminus (spectacles without overminus or no spectacles) in children with intermittent exotropia (IXT) 3 to <7 years of age is to determine whether to proceed to a full-scale, longer-term randomized trial.

DETAILED DESCRIPTION:
The objective of this short-term, pilot randomized trial comparing 2.50D overminus lens treatment vs. non-overminus (spectacles without overminus or no spectacles) is to determine whether to proceed to a full-scale, longer-term randomized trial. This decision will be based primarily on assessing the initial (8-week) response to overminus by comparing treatment groups on the following outcomes:

* Mean distance IXT control score (each patient's score is the mean of 3 control scores) (primary outcome)
* The proportion of subjects with treatment response, defined as 1 or more points improvement in mean of 3 distance IXT control scores (secondary outcome)
* Adverse effects, near visual acuity outcomes, and spectacle wear compliance

ELIGIBILITY:
The following criteria must be met for the child to be enrolled in the study:

* Age 3 years to < 7 years
* Intermittent exotropia (manifest deviation) meeting all of the following criteria:

  * Intermittent exotropia or constant exotropia at distance

    * Mean distance control score of 2 points or more (mean of 3 assessments over the exam)
  * Intermittent exotropia, exophoria, or orthophoria at near

    * Subject cannot have a score of 5 points on all 3 near assessments of control
  * Exodeviation at least 15∆ at distance measured by PACT
  * Near deviation does not exceed distance deviation by more than 10∆ by PACT (convergence insufficiency type IXT excluded)
* No previous non-surgical treatment for IXT (other than refractive correction), including vision therapy for IXT, within the past 6 months.
* No previous substantial overminus treatment, defined as wearing spectacles that are overminused by 1.00D SE or more (treatment with lenses overminused by less than 1.00D SE is allowed at any time prior to enrollment).
* No vision therapy, patching, atropine, or other penalization for amblyopia during the last 2 weeks
* No prior strabismus, intraocular, or refractive surgery (including BOTOX injection)
* Cycloplegic refraction within 7 months, but NOT on the day of enrollment
* Spherical equivalent (SE) in both eyes between -6.00D and +1.00D inclusive
* Distance visual acuity 0.3 logMAR (20/40) or better (by ATS-HOTV) in both eyes
* No interocular difference of distance visual acuity more than 0.2 logMAR (2 lines)
* Child must be wearing refractive correction (pre-study spectacles) for at least 1 week if refractive error (based on cycloplegic refraction performed within 7 months) meets any of the following:

  * SE anisometropia ≥1.00 D
  * Astigmatism ≥1.00 D in either eye
  * SE myopia ≥-0.50 D in either eye
* Refractive correction must meet the following criteria relative to the cycloplegic refraction:

  * SE anisometropia must be within <1.0D of the SE anisometropic difference
  * Astigmatism must be within <1.00D of full magnitude; axis must be within 10 degrees if ≤1.00D, and within 5 degrees if >1.00D.
  * The SE of the spectacles must be within <1.00D of the full cycloplegic refraction SE.

    * A correction that yields at least 1.00 D more minus SE than the cycloplegic refraction SE is considered previous substantial overminus lens treatment and the patient is not eligible.
* No current contact lens wear
* No abnormality of the cornea, lens, or central retina
* Gestational age ≥ 32 weeks
* Birth weight > 1500 grams
* No Down syndrome or cerebral palsy
* No severe developmental delay which would interfere with treatment or evaluation (in the opinion of the investigator). Subjects with mild speech delays or reading and/or learning disabilities are not excluded.
* No disease known to affect accommodation, vergence, and ocular motility such as multiple sclerosis, Graves orbitopathy, myasthenia gravis, diabetes mellitus, or Parkinson disease
* No current use of any ocular or systemic medication known to affect accommodation or vergence, such as anti-anxiety agents (e.g., Librium or Valium), anti-arrhythmic agents (e.g., Cifenline, Cibenzoline), anti-cholinergics (e.g., motion sickness patch (scopolamine)), bladder spasmolytic drugs (e.g., Propiverine), hydroxychloroquine, chloroquine, phenothiazines (e.g., Compazine, Mellaril, Thorazine), tricyclic antidepressants (e.g., Elavil, Nortriptyline, Tofranil)
* Parent understands the protocol and is willing to accept randomization to overminus spectacles or non-overminus status
* Parent has home phone (or access to phone) and is willing to be contacted by Jaeb Center staff and Investigator's site staff
* Relocation outside of area of an active PEDIG site within next 8 weeks is not anticipated

Ages: 3 Years to 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 58 (Actual)
Dates: Start 2014-12; Primary Completion 2015-07 (Actual); Study Completion 2015-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan M Holmes, MD, Study Chair — Mayo Clinic; Angela M Chen, OD, MS, Study Chair — Marshall B. Ketchum University
Locations (2):
- United States (2):
  - Marshall B. Ketchum University, Fullerton, California
  - Mayo Clinic, Rochester, Minnesota

IPD SHARING:
Plan to Share IPD: Yes
In accordance with the NIH data sharing policy, a de-identified database is placed in the public domain on the PEDIG public website after the completion of each protocol and publication of the primary manuscript.

REFERENCES:
- [Result] Pediatric Eye Disease Investigator Group; Chen AM, Holmes JM, Chandler DL, Patel RA, Gray ME, Erzurum SA, Wallace DK, Kraker RT, Jensen AA. A Randomized Trial Evaluating Short-term Effectiveness of Overminus Lenses in Children 3 to 6 Years of Age with Intermittent Exotropia. Ophthalmology. 2016 Oct;123(10):2127-36. doi: 10.1016/j.ophtha.2016.06.042. Epub 2016 Aug 6. PMID 27506485
- See also: PEDIG Public Website — http://pedig.jaeb.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Between December 2014 and May 2015, 58 children were enrolled at 21 sites, with 31 participants assigned to observation and 27 to overminus treatment.
Period: Overall Study
Arm/Group | Overminus Treatment | Non-overminus Treatment
Started | 27 | 31
Completed | 27 | 31
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Overminus Treatment | Non-overminus Treatment | Total
Number analyzed (Participants) | 27 | 31 | 58
Age, Continuous [Mean (Standard Deviation); unit: years] | 5.2 (1) | 5.1 (1.2) | 5.1 (1.1)
Age, Customized [Number; unit: participants] — Baseline age reflects age at randomization. The age eligibility requirement at enrollment was 3 to <7 years old.
  participants
    3 to <4 years | 7 | 3 | 10
    4 to <5 years | 4 | 11 | 15
    5 to <6 years | 9 | 10 | 19
    6 to <7 years | 7 | 7 | 14
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18 | 18 | 36
  Male | 9 | 13 | 22
Race/Ethnicity, Customized [Number; unit: participants]
  White | 14 | 15 | 29
  Black/African American | 2 | 4 | 6
  Hispanic or Latino | 6 | 9 | 15
  Asian | 5 | 3 | 8
Refractive error in more myopic eye (spherical equivalent, D) [Number; unit: participants]
  >+0.50 to +1.00 | 13 | 15 | 28
  0 to +0.50 | 5 | 9 | 14
  <0 to >-0.50 | 2 | 1 | 3
  -0.50 to >-1.00 | 4 | 1 | 5
  -1.00 to >-1.50 | 1 | 0 | 1
  -1.50 to >-2.00 | 1 | 0 | 1
  -2.00 to >-2.50 | 0 | 2 | 2
  -2.50 to >-3.00 | 0 | 2 | 2
  <=-3.00 | 1 | 1 | 2
Accommodative convergence over accommodation (AC/A) ratio [Number; unit: participants] — Accommodative convergence over accommodation (AC/A) ratio calculated by taking the difference between the distance (6m) Prism Alternate Cover Test measurements with the participant wearing habitual correction and with the participant wearing -2.00D lenses over the habitual correction, and dividing the difference by 2.
  participants
    <2.5 | 12 | 13 | 25
    2.5 to 6.0 | 12 | 15 | 27
    >6.0 | 3 | 3 | 6

OUTCOME MEASURES:

1. Primary Outcome: Mean Distance Exotropia Control Score
Description: At each visit, control of the exodeviation was measured at distance (6 meters) and at near (1/3 meters) using the Office Control Score* which ranges from 0 (phoria, best control) to 5 (constant exotropia, worst control). Due to the variability of single measures of control, we used a "triple control score," which is a mean of 3 measures obtained at specific time-points during a 20- to 40-minute office examination. The primary analysis was an intention-to-treat treatment group comparison of mean 8-week distance control using an analysis of covariance (ANCOVA) model which adjusted for baseline distance control.
  *Mohney BG, Holmes JM. An office-based scale for assessing control in intermittent exotropia. Strabismus 2006;14(3):147-50.
Time Frame: 8 weeks
Measure: Mean (Standard Deviation); unit: points on control score scale
Arm/Group | Overminus Treatment | Non-overminus Treatment
Number analyzed (Participants) | 27 | 31
points on control score scale | 2.0 (1.4) | 2.8 (1.4)
Statistical Analysis 1: Comparison: Overminus Treatment vs Non-overminus Treatment; Test type: Superiority or Other; p = 0.01, ANCOVA — P-value is calculated for one-sided hypothesis test; Comparison of mean 8-wk distance control using ANCOVA adjusted for baseline distance control pre-study spectacle wear, and pre-study IXT treatment; Mean Difference (Final Values) = -0.75, 95% CI 2-sided [-1.42 to -0.07] — Difference in mean distance control (overminus - observation) and 95% CI from ANCOVA model adjusting for baseline control, pre-study spectacle wear, and pre-study treatment for IXT. + difference suggests observation group worse than overminus group

2. Secondary Outcome: Mean Near Exotropia Control Score
Description: At each visit, control of the exodeviation was measured at near (1/3 meters) using the Office Control Score which ranges from 0 (phoria, best control) to 5 (constant exotropia, worst control). Due to the variability of single measures of control, we used a "triple control score," which is a mean of 3 measures obtained at specific time-points during a 20- to 40-minute office examination. The secondary analysis was an intention-to-treat treatment group comparison of mean 8-week near control using an analysis of covariance (ANCOVA) model which adjusted for baseline near control.
Time Frame: 8 weeks
Measure: Mean (Standard Deviation); unit: points on control score scale
Arm/Group | Overminus Treatment | Non-overminus Treatment
Number analyzed (Participants) | 27 | 31
points on control score scale | 0.9 (1.2) | 1.2 (1.1)
Statistical Analysis 1: Comparison: Overminus Treatment vs Non-overminus Treatment; Test type: Superiority or Other; p = 0.14, ANCOVA — P-value is calculated for one-sided hypothesis test; Comparison of mean 8-wk near control using ANCOVA adjusted for baseline near control pre-study spectacle wear, and pre-study IXT treatment; Mean Difference (Final Values) = -0.24, 95% CI 2-sided [-0.68 to 0.19] — Comparison of mean 8-wk distance control using ANCOVA adjusted for baseline near control pre-study spectacle wear, and pre-study IXT treatment

3. Secondary Outcome: Distribution of Distance Control Score at 8-week Outcome
Description: Control of exodeviation will be assessed in the habitual correction at distance (6 meters) and near (1/3 meter) using a standardized IXT control scale.
Time Frame: 8 weeks
Measure: Number; unit: participants
Arm/Group | Overminus Treatment | Non-overminus Treatment
Number analyzed (Participants) | 27 | 31
participants
  0 to <1 | 4 | 1
  1 to <2 | 11 | 7
  2 to <3 | 5 | 10
  3 to <4 | 1 | 3
  4 to 5 | 6 | 10

4. Secondary Outcome: Distribution of Near Control Score at 8-week Outcome
Description: as for outcome 3
Time Frame: 8 weeks
Measure: Number; unit: participants
Arm/Group | Overminus Treatment | Non-overminus Treatment
Number analyzed (Participants) | 27 | 31
participants
  0 to <1 | 15 | 10
  1 to <2 | 7 | 13
  2 to <3 | 2 | 3
  3 to <4 | 2 | 5
  4 to 5 | 1 | 0

5. Secondary Outcome: Proportion of Subjects With Distance Control Treatment Response
Description: A comparison of the proportion of subjects showing a "treatment response," defined as an improvement of at least 1 point in distance control (mean of the 3 assessments over the exam) between enrollment and 8 weeks.
Time Frame: 8 weeks
Measure: Number; unit: participants
Arm/Group | Overminus Treatment | Non-overminus Treatment
Number analyzed (Participants) | 27 | 31
participants | 16 | 12
Statistical Analysis 1: Comparison: Overminus Treatment vs Non-overminus Treatment; Test type: Superiority or Other; p = 0.07, Chi-squared — The p-value was not adjusted for multiple comparisons; Risk Difference (RD) = 21, 95% CI 2-sided [-6 to 45]

6. Secondary Outcome: Symptom Survey Response to Question: Has Child Looked Over His/Her Spectacles Since Enrollment?
Description: A brief survey of symptoms that may be associated with overminus such as headaches, eye strain, and problems with spectacle wear will be administered to the parents of the subjects. Parents are asked to respond to the survey questions based on their observations of their child in the past 2 weeks. Response options are based on frequency of observations; never, rarely, sometimes, often, always, and not applicable. Survey items were derived based on expert opinion of pediatric ophthalmologists and optometrists on the study planning committee. The response options were a 5-point Likert-type scale based on frequency of observations: never = score of 0, almost never = 1, sometimes = 2, often = 3, and always = 4.
Time Frame: 8 weeks
Population: Spectacle-related questions at follow up apply only to observation participants prescribed correction (N=10 (32%) and to all overminus group participants N=27 (100%)).
Measure: Number; unit: participants
Groups:
- Overminus Treatment: Spectacle-related questions at follow up apply to all overminus group participants.
- Non-overminus Treatment: Spectacle-related questions at follow up apply only to non-overminus group participants prescribed correction spectacles.
Arm/Group | Overminus Treatment | Non-overminus Treatment
Number analyzed (Participants) | 27 | 10
participants
  Looked over specatcles: Always | 0 | 0
  Looked over specatcles: Often | 3 | 1
  Looked over specatcles: Sometimes | 7 | 2
  Looked over specatcles: Rarely | 2 | 2
  Looked over specatcles: Never | 15 | 5

7. Secondary Outcome: Stereoacuity
Description: Stereoacuity will be assessed with habitual correction using the Randot Preschool stereotest at near (performed at 40 cm). A specific level of stereoacuity is not required for eligibility.
Time Frame: 8 weeks
Measure: Mean (Standard Deviation); unit: log arcsecond
Arm/Group | Overminus Treatment | Non-overminus Treatment
Number analyzed (Participants) | 27 | 31
log arcsecond | 2.2 (0.5) | 2.2 (0.6)

8. Secondary Outcome: Distance Visual Acuity
Description: Monocular distance visual acuity testing with the habitual correction and without cycloplegia was measured using the Amblyopia Treatment Study HOTV testing protocol on any certified visual acuity system. The treatment groups were not different with respect to 8-week control PACT at distance
Time Frame: 8 weeks
Measure: Mean (Standard Deviation); unit: prism diopters
Arm/Group | Overminus Treatment | Non-overminus Treatment
Number analyzed (Participants) | 27 | 31
prism diopters | 21.1 (11.2) | 23.0 (6.3)

9. Secondary Outcome: Binocular Near Visual Acuity
Description: Binocular near visual acuity was tested in habitual correction using the ATS4 near visual acuity test. The treatment groups were not different with respect to 8-week control at near.
Time Frame: 8 weeks
Measure: Mean (Standard Deviation); unit: prism diopters
Arm/Group | Overminus Treatment | Non-overminus Treatment
Number analyzed (Participants) | 27 | 31
prism diopters | 12.8 (8.3) | 16.9 (8.4)

10. Secondary Outcome: Symptom Survey Response to Question: Has Your Child Had Eyestrain (Tired, Sore, or Uncomfortable Eyes)?
Description: as for outcome 6
Time Frame: 8 weeks
Measure: Number; unit: participants
Arm/Group | Overminus Treatment | Non-overminus Treatment
Number analyzed (Participants) | 27 | 31
participants
  Always | 0 | 0
  Often | 0 | 0
  Sometimes | 4 | 3
  Rarely | 5 | 4
  Never | 18 | 24

11. Secondary Outcome: Symptom Survey Response to Question: Since Enrollment Has Your Child Avoided Reading or Doing Things up Close?
Description: as for outcome 6
Time Frame: 8 weeks
Population: as for outcome 6
Measure: Number; unit: participants
Arm/Group | Overminus Treatment | Non-overminus Treatment
Number analyzed (Participants) | 27 | 31
participants
  Always | 0 | 0
  Often | 0 | 0
  Sometimes | 1 | 1
  Rarely | 0 | 2
  Never | 26 | 28

12. Secondary Outcome: Symptom Survey Response to Question: Has Your Child Reported Blurry Vision?
Description: as for outcome 6
Time Frame: 8 weeks
Measure: Number; unit: participants
Arm/Group | Overminus Treatment | Non-overminus Treatment
Number analyzed (Participants) | 27 | 31
participants
  Always | 0 | 0
  Often | 0 | 0
  Sometimes | 1 | 1
  Rarely | 1 | 1
  Never | 25 | 29

13. Secondary Outcome: Proportion of Subjects With Near Control Treatment Response
Description: A comparison of the proportion of subjects showing a "treatment response," defined as an improvement of at least 1 point in near control (mean of the 3 assessments over the exam) between enrollment and 8 weeks.
Time Frame: 8 weeks
Measure: Number; unit: participants
Arm/Group | Overminus Treatment | Non-overminus Treatment
Number analyzed (Participants) | 27 | 31
participants | 7 | 8
Statistical Analysis 1: Comparison: Overminus Treatment vs Non-overminus Treatment; Test type: Superiority or Other; p = 0.54, Chi-squared — The p-value was not adjusted for multiple comparisons; Risk Difference (RD) = 0.001, 95% CI 2-sided [-23 to 24]

ADVERSE EVENTS:
Time Frame: Baseline to 8 weeks after randomization.
Arm/Group | Overminus Treatment | Non-overminus Treatment
Serious Adverse Events (participants affected / at risk) | 0/27 | 0/31
Other Adverse Events (participants affected / at risk) | 3/27 | 2/31
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Overminus Treatment (N=27) | Non-overminus Treatment (N=31)
Development of esodeviation (Eye disorders) | 1 (1) | 0 (0) — One participant had near deviation change from 12 PD exodeviation at baseline to 3 PD esodeviation at 8 weeks. During same period, exodeviation at distance changed from 20 PD to 12 PD and stereoacuity at near changed from 100 arcsec to 60 arcsec.
Reduction in monocular distance visual acuity >=2 lines (Eye disorders) | 2 (2) | 1 (1)
Reduction in binocular near visual acuity >=2 lines (Eye disorders) | 0 (0) | 1 (1)

LIMITATIONS AND CAVEATS:
Small sample size; only 8-weeks of follow up; high test-retest variability of control; some regression to the mean may be present; do not know if treatment effect would persist after overminus lenses are replaced with usual spectacle correction.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No